CLINICAL TRIAL: NCT00388089
Title: Phase I Study of Weekly Bortezomib (VELCADE, PS-341) and Weekly Topotecan (HYCAMTIN) in Solid Tumor Patients With an Emphasis on Small Cell Lung Cancer (SCLC)
Brief Title: Bortezomib and Topotecan in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Angela Davies, MD, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000505990; P30CA093373 (NIH); UCDCC-157 (Other: University of California, Davis - Cancer Center); 200412738 (Other: University of California, Davis - IRB); GSK-8531 (Other Grant/Funding Number: GlaxoSmithKline); MILLENNIUM-X05131 (Other Grant/Funding Number: Millennium Pharmaceuticals)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2007-12

CONDITIONS: Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Bortezomib; Topotecan; Flow Cytometry; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bortezomib — Dose level A: 1 mg/m2; Dose level B: 1.3 mg/m2; Dose level C: 1.6 mg/m2; Dose level D: 1.6 mg/m2
  Other Names: PS-341, Velcade
Drug: topotecan hydrochloride — Dose level A: 3 mg/m2; Dose level B: 3 mg/m2; Dose level C: 3 mg/m2; Dose level D: 4 mg/m2
  Other Names: Hycamtin
Other: flow cytometry — No description
Other: immunoenzyme technique — No description
Other: immunohistochemistry staining method — No description
Other: laboratory biomarker analysis — No description

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with topotecan may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib and topotecan in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and feasibility of bortezomib and topotecan hydrochloride in patients with advanced solid tumors.

Secondary

* Determine the maximum tolerated dose (MTD) of bortezomib and topotecan hydrochloride in these patients.
* Determine, preliminarily, the efficacy of this regimen in these patients.
* Perform laboratory correlative studies on tumor tissue and blood samples from these patients to investigate potential predictors of response.
* Obtain fresh tumor tissue for correlative studies from a subset of patients with small cell lung cancer treated at the MTD.

OUTLINE: This is a dose-escalation study.

Patients receive topotecan hydrochloride IV over 30 minutes followed by bortezomib IV on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may continue to receive bortezomib alone in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan hydrochloride and bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Ten additional patients with small cell lung cancer are treated at the MTD. These patients undergo tumor biopsy at baseline and before the second course of therapy.

Tumor tissue is collected at baseline in all patients. Blood samples are collected at baseline, at the beginning of courses 2 and 3, and after completion of study treatment. Samples are examined for topoisomerase-1 levels by western blotting; BCL-2, BCL-xL, BAX, and p27 by immunohistochemistry; hypoxia-inducible factor-1, plasminogen-activator inhibitor 1, vascular endothelial growth factor, and osteopontin by immunoenzyme techniques; and NF-kB and p27 nuclear expression by flow cytometry.

After completion of study treatment, patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor, meeting 1 of the following criteria:

  * Disease progressed after ≥ 1 prior standard therapy regimen
  * Treatment-naive with no standard therapy of curative intent available
  * Not a candidate for standard therapy due to poor performance status
* Patients with small cell lung cancer are enrolled after the maximum tolerated dose has been determined

  * Must have tumor accessible for biopsy
* Measurable disease by RECIST criteria or evaluable disease (e.g., pleural effusion, ascites, or bone metastasis)

  * Disease in previously irradiated sites is considered measurable provided there is clear disease progression after radiotherapy
* Asymptomatic brain metastasis treated by prior surgical resection or radiotherapy allowed if both of the following criteria are met:

  * Neurologically stable
  * Off steroids and anticonvulsants for ≥ 4 weeks

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine clearance ≥ 40 mL/min
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3.0 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No preexisting neuropathy ≥ grade 2 within the past 14 days
* No hypersensitivity to bortezomib, boron, or mannitol
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina, severe uncontrolled ventricular arrhythmias, or ECG evidence of acute ischemia or active conduction system abnormalities

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Any number of prior chemotherapy regimens allowed
* At least 4 weeks since prior chemotherapy and recovered
* At least 2 weeks since prior radiotherapy and recovered
* No prior topotecan hydrochloride or bevacizumab
* At least 14 days since prior investigational drugs
* No concurrent anticonvulsants metabolized by the cytochrome P450 pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety | Monitored on an ongoing basis during the study
  If cumulative toxicities are seen in subsequent treatment cycles, a decision regarding modification or discontinuation of the study drug and/or patient enrollment will be made by the sponsor in conjunction with the investigator.

SECONDARY OUTCOMES:
Toxicity | On Day 8 and at beginning of subsequent cycles
  Toxicity will be evaluated based on the standard NCI CTC grading criteria version 3.0.
Response rate | At baseline and every 2 courses during treatment
  As assessed by RECIST criteria
Best response | From start of treatment until disease progression/recurrence
  Best response is determined from the sequence of objective status.
Survival | From registration to time of death due to any cause
  Patients will be followed for 30 days after removal from study treatment or until all treatment-related toxicities resolve to < grade 1.
Progression-free survival | From registration to the first observation of disease progression or death due to any cause
  If a patient has not progressed or died, progression-free survival is censored at the time of last follow-up.
Topoisomerase levels as assessed by western blot and tumor tissue biopsy | From pre-treatment to post-treatment
  The aim of these molecular correlates is to examine the relationship between these studies and the clinical response to treatment.
NF-kB and BCL-2 family activity as assessed by immunohistochemistry | From pre-treatment to post-treatment
  The aim of these molecular correlates is to examine the relationship between these studies and the clinical response to treatment.
Loss of p27 as assessed by immunohistochemistry | From pre-treatment to post-treatment
  The aim of these molecular correlates is to examine the relationship between these studies and the clinical response to treatment.
Hypoxia-induced plasma proteins as measured by enzyme-linked immunosorbent assay (ELISA) | From pre-treatment to post-treatment
  The aim of these molecular correlates is to examine the relationship between these studies and the clinical response to treatment.
Shed tumor DNA in plasma | From pre-treatment to post-treatment
  The aim of these molecular correlates is to examine the relationship between these studies and the clinical response to treatment.
Biological activity of bortezomib as measured by flow cytometry | From pre-treatment to post-treatment
  The aim of these molecular correlates is to examine the relationship between these studies and the clinical response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Davies, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States